CLINICAL TRIAL: NCT01062165
Title: Population Pharmacokinetic Analysis of Caspofungin in Overweight and Obese Volunteers
Brief Title: Effect of Weight and/or Obesity on Caspofungin Drug Concentrations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ron Hall, Associate Professor, Texas Tech University Health Sciences Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TTHSC-A09-3566; 5UL1RR024982-02 (NIH)
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Obesity; Fungal Infection
Keywords: Echinocandin; Obesity; Pharmacokinetics; Pharmacodynamics; Fungal infection
MeSH Terms: conditions — Obesity; Mycoses | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capsofungin (Experimental): Six volunteers will have a body mass index (BMI) less than 25 kg/m2, 6 will have a BMI 25-40 kg/m2, and 6 will have a BMI greater than 40 kg/m2.
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — Caspofungin 70mg IV (each volunteer will only receive one dose of the study drug)
  Other Names: Cancidas

SUMMARY:
This study will find how weight affects the dosing of a drug called caspofungin. Currently, the amount of caspofungin a patient receives is the same regardless of the patient's weight.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 18 years of age or older, of all racial and ethnic origins. English and/or Spanish speaking volunteers are eligible to participate.

Exclusion Criteria:

* Pregnant or nursing or unwilling to use a reliable contraception method during the study. The effects of caspofungin on pregnancy are unknown. In addition, the metabolic changes that accompany pregnancy may alter the concentration-time profile of caspofungin, so that the pregnancy and post-partum state would be a confounding variable.
* Abnormal liver function tests: transaminases>10 times upper limit of normal, Alkaline phosphatase>5 times upper limit of normal, total bilirubin>5 times upper limit of normal.
* History of allergies to echinocandins.
* Echinocandins are contraindicated for any reason.
* Volunteers unwilling to comply with study procedures.
* Suspected or documented systemic fungal infection.
* Concomitant use of rifamycins, tacrolimus, or cyclosporine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hall, PharmD, MSCS, Principal Investigator — Texas Tech University HSC
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Result] Hall RG 2nd, Swancutt MA, Meek C, Leff R, Gumbo T. Weight drives caspofungin pharmacokinetic variability in overweight and obese people: fractal power signatures beyond two-thirds or three-fourths. Antimicrob Agents Chemother. 2013 May;57(5):2259-64. doi: 10.1128/AAC.01490-12. Epub 2013 Mar 4. PMID 23459494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers recruited with fliers at medical center.
Groups:
- Capsofungin: Six volunteers will have a body mass index (BMI) less than 25 kg/m2, 6 will have a BMI 25-40 kg/m2, and 6 will have a BMI greater than 40 kg/m2.
  Caspofungin : Caspofungin 70mg IV (each volunteer will only receive one dose of the study drug)
Period: Overall Study
Arm/Group | Capsofungin
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Capsofungin
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (13.2)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Total Clearance of Caspofungin
Time Frame: 0-72 hours (0, 1, 8, 16, 24, 48, and 72 hours)
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Capsofungin
Number analyzed (Participants) | 18
L/hr | 0.508 (0.223)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Capsofungin
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capsofungin (N=18)
Headache (General disorders) | 1 (1) — Classified as mild by the investigators. Resolved about 30 minutes after 650 mg of acteminophen was administered. Volunteer had a history of headaches and migraines.
Hot flashes and sweating (General disorders) | 1 (1) — Symptoms resolved within a few hours without any intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No